CLINICAL TRIAL: NCT03879538
Title: A Prospective Randomized Controlled Pilot Study Nitrous Oxide for the Treatment of Complex Regional Pain Syndrome
Brief Title: Nitrous Oxide for the Treatment of Complex Regional Pain Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-150
Record Dates: First submitted 2019-01-31; First posted 2019-03-18 (Actual); Results first posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Complex Regional Pain Syndrome
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Nitrous Oxide; Oxygen

STUDY DESIGN:
Intervention Model Description: The nitrous oxide group will receive 50% nitrous oxide mixed with 50% oxygen, and the control group will receive 50% oxygen (oxygen plus air mixture). Both groups will undergo inhalation therapy for a duration of 2 hours via an FDA-approved mask breathing circuit. Vital signs (blood pressure, respiratory rate, heart rate) will be monitored every 30 minutes.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and other involved providers will be blinded to the treatment type. Research investigators administering the treatments will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- The nitrous oxide group (Active Comparator): Nitrous oxide group will receive 50% nitrous oxide mixed with 50% oxygen, inhalation therapy for a duration of 2 hours via an FDA-approved mask breathing circuit.
  Interventions: Drug: Nitrous Oxide
- The Control Group (Placebo Comparator): Control group will receive 50% oxygen, inhalation therapy for a duration of 2 hours via an FDA-approved mask breathing circuit.
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Nitrous Oxide — A total of three inhalation treatments with 50% Nitrous Oxide plus 50% oxygen (6 total exposure hours) over one week with 2 or 3 days between each session.
  Other Names: 50 % Nitrous Oxide plus 50% Oxygen
  Arms: The nitrous oxide group
Drug: Oxygen — A total of three inhalation treatments with 50% oxygen (6 total exposure hours) over one week with 2 or 3 days between each session.
  Other Names: 50% Oxygen
  Arms: The Control Group

SUMMARY:
Patients will then be randomized via a web-based randomization system Redcap Allocation will be stratified based on the presence of a pre-existing spinal cord stimulator to either the nitrous oxide study group or the oxygen control group.

The nitrous oxide group will receive 50% nitrous oxide mixed with 50% oxygen, and the control group will receive 50% oxygen (oxygen plus air mixture). Both groups will undergo inhalation therapy for a duration of 2 hours via an FDA-approved mask breathing circuit. Vital signs (blood pressure, respiratory rate, heart rate) will be monitored every 30 minutes. Pulse oximetry monitoring will be continuous. Patients will be monitored for side effects including nausea, vomiting, desaturation, sedation, respiratory depression, and dizziness. Patients and other involved providers will be blinded to the treatment type.

DETAILED DESCRIPTION:
Daily opioid consumption data will be collected by having patients record and report their daily opioid use before and after treatment. Oral and transdermal opioids will be converted to standardized morphine equivalents and adjusted for bioavailability.

Patients will present for the first scheduled treatment and they will fill out the PROMIS-29 v2 survey and the SF-MPQ-2 (6 neuropathic pain items). Patients will also turn in their opioid use log.

Vital signs will be obtained. Patients with significantly abnormal vital signs or vital signs that are significantly deviated from baseline will be referred to appropriate medical care.

Patients will then be randomized via a web-based randomization system Redcap. Group allocation will be stratified based on the presence of a pre-existing spinal cord stimulator to either the nitrous oxide study group or the oxygen control group.

The nitrous oxide group will receive 50% nitrous oxide mixed with 50% oxygen, and the control group will receive 50% oxygen. Both groups will undergo inhalation therapy for a duration of 2 hours via an FDA-approved mask breathing circuit. Active Control, because patients may be able to tell if they are receiving nitrous oxide, patient blinding may be compromised. Therefore, we plan to utilize an active control. Both groups will receive 2 mg of intravenous midazolam, to infuse over 5 minutes, at the start of each breathing treatment session. IVs will be removed at the conclusion of each breathing treatment. Vital signs (blood pressure, respiratory rate, heart rate) will be monitored every 30 minutes. Pulse oximetry monitoring will be continuous. Patients will be monitored for side effects including nausea, vomiting, desaturation, sedation, respiratory depression, and dizziness. Patients and other involved providers will be blinded to the treatment type. Research investigators administering the treatments will not be blinded.

At the conclusion of inhalation therapy, the gas will be turned off and patients will breathe room air. All patients will be monitored for an additional 30 minutes. This recovery time is more than sufficient to ensure nitrous oxide is completely eliminated in those patients who receive it. Patients will be monitored and asked about side effects.

Patients will receive a total of three treatments (6 total exposure hours) over one week with 2 or 3 days between each session. Possible treatment schedules: Monday-Wednesday-Friday, Wednesday-Friday-Monday, or Friday-Monday-Wednesday. After the conclusion of the third treatment, patients will be followed with phone calls as detailed in the Measurement section below.

1. Drug Handling Instructions

a. Nitrous oxide for the study will be stored at room temperature in appropriately labeled E-cylinder tanks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be diagnosed with CRPS based on the revised International Association for the Study of Pain criteria.
2. Duration of disease must be at least 6 months.
3. Written informed consent.

Exclusion Criteria:

1. Patients who had no subjective benefit from ketamine infusions, as determined by interview during the recruitment process.
2. Patients taking more than 60mg of morphine equivalents or more daily for an alternative chronic pain condition.
3. Patients with both coronary artery disease (as determined by cardiac catheterization) and a functional status of less than 4 metabolic equivalents. The limited functional status must be secondary to cardiopulmonary symptoms (angina, dyspnea on exertion). Patients with coronary artery disease and a limited functional status (<4 METS) secondary to chronic pain can be included.
4. Patients with congestive heart failure of any etiology that are NYHA Class III or IV
5. Patients with moderate or severe pulmonary hypertension as determined by echocardiogram or right heart catheterization.
6. Patients with intraocular surgery within the past 14 days
7. Patients with worker's compensation claims and active litigation.
8. Patients who have been diagnosed with COPD.
9. Patients who use home oxygen therapy for any condition.
10. Diagnosis of Alcohol Use Disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
11. Illicit drug use within the past three months (not including marijuana).
12. Pregnant patients or patients with upcoming planned pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hale, MD, Principal Investigator — Anesthesiologist
Locations (1):
- Cleveland Clinic Pain Management, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- The Control Group: Control group will receive 100% oxygen, inhalation therapy for a duration of 2 hours via an FDA-approved mask breathing circuit.
  Oxygen: A total of three inhalation treatments with 100% oxygen (6 total exposure hours) over one week with 2 or 3 days between each session.
Period: Overall Study
Arm/Group | The Nitrous Oxide Group | The Control Group
Started | 20 | 24
Completed | 20 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The Nitrous Oxide Group | The Control Group | Total
Number analyzed (Participants) | 20 | 24 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (12.3) | 46.3 (13.4) | 45.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 22 | 38
  Male | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian | 20 | 21 | 41
  Race: Black/African American | 0 | 1 | 1
  Race: Hispanic/Latino | 0 | 1 | 1
  Race: Multicultural | 0 | 1 | 1
Duration of disease [Median (Inter-Quartile Range); unit: months] | 53.5 [36.5 to 126.0] | 108.0 [28.5 to 122.5] | 89.5 [32.0 to 122.5]
Spinal cord stimulators used [Count of Participants; unit: Participants] | 5 | 7 | 12
Extremity affected [Count of Participants; unit: Participants]
  Single location | 8 | 5 | 13
  Multiple locations | 12 | 19 | 31
Pain score at baseline [Mean (Standard Deviation); unit: units on a scale] — Patients-reported pain score was the item 29 in PROMIS-29 Profile v2.0, with scales ranging from 0 - 'no pain' to 10 - 'worst pain ever'.
  units on a scale | 7.3 (1.7) | 6.8 (1.5) | 7.0 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: scales ranging from 0 - "no pain" to 10 - "worst pain ever" based on the PROMIS-29 v2.0 questionnaire.
Time Frame: one-week and one-month follow-up time points
Population: A few patients had missing primary outcome measurements. The Mean (SD) values presented here was based on available raw data. In our formal analysis of treatment effect on primary outcome, we used multiple imputation procedures to impute missing primary outcome values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Nitrous Oxide Group | The Control Group
Number analyzed (Participants) | 20 | 24
score on a scale
  one-week follow-up: number analyzed (Participants) | 19 | 23
  one-week follow-up | 5.9 (1.5) | 6.0 (2.5)
  one-month follow-up: number analyzed (Participants) | 17 | 21
  one-month follow-up | 6.5 (2.0) | 6.8 (2.2)
Statistical Analysis 1: Comparison: The Nitrous Oxide Group vs The Control Group; Null hypothesis: Mean of pain score assessed at one-week and one-month follow-up after end of treatment for Nitrous Oxide group equals that assessed at same time points for the Control group; Test type: Superiority; p = 0.19, Mixed Models Analysis — a priori threshold for statistical significance was p = 0.05; Mean Difference (Net) = -0.57, 95% CI 2-sided [-1.42 to 0.28] — Mean difference is Nitrous Oxide minus Control

2. Secondary Outcome: PROMIS-29 Survey Physical Health Z-score, Mental Health Z-score
Description: As intermediate scores, T-scores for each of the 7 domains used in the survey need to be estimated from raw data in order to obtain final summary Z-scores measuring physical and mental health. T-scores were obtained from an on-line service provided by the HealthMeasures Scoring Service (https://www.assessmentcenter.net/ac_scoringservice). Physical and mental summary Z-scores were calculated using the formulas given in the document titled "Calculating physical and mental health summary scores for PROMIS-29 v2.0 and v2.1" (dated on August 8, 2018) by Karen L. Spritzer and Ron D. Hays from the website HealthMeasures.net.
  High T-scores indicates more of the concept being measured which can be either desirable or undesirable outcome, e.g., high T-score on fatigue is undesirable whereas desirable for physical function. Z-scores are standard scores with mean of 0 and SD of 1 in reference population. High Z-scores are desirable for either physical or mental health.
Time Frame: one-week and one-month follow-ups after treatments were ended
Population: A few patients had missing values due to withdrawal from the study or failure of follow-up contact.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | The Nitrous Oxide Group | The Control Group
Number analyzed (Participants) | 20 | 24
z-score
  Physical health Z-score at one-week follow-up: number analyzed (Participants) | 19 | 23
  Physical health Z-score at one-week follow-up | -1.4 (0.71) | -1.4 (0.78)
  Physical health Z-score at one-month follow-up: number analyzed (Participants) | 17 | 21
  Physical health Z-score at one-month follow-up | -1.4 (0.58) | -1.5 (0.68)
  Mental health Z-score at one-week follow-up: number analyzed (Participants) | 19 | 23
  Mental health Z-score at one-week follow-up | -1.01 (0.81) | -0.91 (1.00)
  Mental health Z-score at one-month follow-up: number analyzed (Participants) | 17 | 21
  Mental health Z-score at one-month follow-up | -1.2 (0.88) | -1.1 (0.91)
Statistical Analysis 1: Comparison: The Nitrous Oxide Group vs The Control Group; Null hypothesis for testing difference in means of physical health Z-score between two study groups: mean of physical health Z-score assessed at one-week and one-month follow-ups for Nitrous Oxide group was equal to that assessed at the same follow-up time points for Control group; Test type: Superiority; p = 0.36, Mixed Models Analysis — a priori threshold for statistical significance is p<0.05; Mean Difference (Net) = 0.13, 95% CI 2-sided [-0.16 to 0.43] — Mean difference is Nitrous oxide minus control
Statistical Analysis 2: Comparison: The Nitrous Oxide Group vs The Control Group; Null hypothesis for testing difference in means of mental health Z-score between two study groups: mean of mental health Z-score assessed at one-week and one-month follow-ups for Nitrous Oxide group was equal to that assessed at the same follow-up time points for Control group; Test type: Superiority; p = 0.66, Mixed Models Analysis — a priori threshold for statistical significance is p<0.05; Mean Difference (Net) = 0.087, 95% CI 2-sided [-0.31 to 0.48] — Mean difference is Nitrous oxide minus control

3. Secondary Outcome: PGIC Scale
Description: patient disease perception as measured by the Patient's Global Impression of Change (PGIC) survey (a seven-point scale ranging from 1 - "no change or condition has gotten worse" to 7 - "very much improve").
Time Frame: one-week and one-month follow-ups.
Population: A few patients had missing values due to withdrawal from the study or study participants can not be reached for follow-up with phone calls.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | The Nitrous Oxide Group | The Control Group
Number analyzed (Participants) | 20 | 24
score on a scale
  PGIC scale at one-week follow-up: number analyzed (Participants) | 19 | 23
  PGIC scale at one-week follow-up | 2 [1 to 5] | 4 [1 to 5]
  PGIC scale at one-month follow-up: number analyzed (Participants) | 17 | 21
  PGIC scale at one-month follow-up | 2 [1 to 4] | 2 [1 to 5]
Statistical Analysis 1: Comparison: The Nitrous Oxide Group vs The Control Group; Null hypothesis: Mean of PGIC scale assessed at one-week and one-month follow-up time points for Nitrous Oxide patients is equal to that assessed at the same time points for Control patients; Test type: Superiority; p = 0.23, Mixed Models Analysis — a priori threshold for statistical significance is p = 0.05; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.85 to 0.46] — Mean difference is Nitrous Oxide minus Control

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | The Nitrous Oxide Group | The Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/24
Other Adverse Events (participants affected / at risk) | 0/20 | 0/24

LIMITATIONS AND CAVEATS:
limitations include the purely subjective nature of pain which was our primary outcome. Validity of the trial thus depends critically on adequacy of blinding. Because many patients can detect inhaled nitrous oxide, we gave all participants midazolam which has similar effects. But it remains possible that some patients could distinguish nitrous oxide from air, and were thus biased.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT03879538/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT03879538/ICF_001.pdf